CLINICAL TRIAL: NCT05997459
Title: A Single Arm, Phase ll Exploratory Clinical Study of Pemetinib in the Treatment of Advanced Gastric Cancer With FGFR Mutation and Previous Standard Treatment Failure
Brief Title: A Single Arm, Phase II Exploratory Clinical Study of Pemitinib in Advanced Gastric Cancer With Previous Standard Therapy Failure the FGFR Variant
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SL-B2023-124-02
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Locally Advanced Unresectable Gastric Cancer
MeSH Terms: interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental)
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib,13.5mg ,QD,po, 2 weeks / 1 week;Q 3W

SUMMARY:
purpose of research： fundamental purpose:

• To evaluate the effectiveness of pemitinib in patients with advanced gastric cancer who have failed standard therapy with fibroblast growth factor receptor 1-3 (FGFR1-3) variant (including but not limited to FGFR1-3 amplification, rearrangement / fusion, mutation, etc.).

Secondary purpose:

* To evaluate the safety and tolerability of pemitinib in patients with advanced gastric cancer who have previously failed standard therapy with the FGFR1-3 variant: including incidence of adverse events (AEs) and serious adverse events (SAEs) and association with therapy. Incidence of treatment-related AEs / SAEs.
* Exploring efficacy and safety in subjects with different FGFR variant types.

The end of the study:

Main end point:

• The primary endpoint of the study was the 6-month PFS rate (progression-free survival, defined as first dose to disease progression [PD] or death).

Secondary end point:

• Objective response rate (defined as the proportion of subjects achieving complete response (CR) or partial response (PR) by RECIST1.1 criteria).

Duration of response (DOR, defined as the time from first CR or PR to PD, is used only for subjects with an objective response).

* Disease control rate (DCR, defined as the proportion of subjects with CR + PR + stable disease stable [SD]).
* Overall survival (OS, defined as the time of first dose to death from any cause).
* Safety and tolerability: Grade evaluation for assessing the severity of adverse events according to NCI CTCAE (version 5.0), including:

  1. Incidence, severity, and association of all AEs, TRAEs, SAEs, and the study drug;
  2. Number and proportion of subjects stopping treatment due to the above adverse events;
  3. Study changes in vital signs, physical examination findings, and laboratory results before, during and after treatment.
* To describe the efficacy and safety in subjects with different FGFR gene variant types.

DETAILED DESCRIPTION:
research design: This study is a prospective, single-arm, phase II clinical study. Patients with advanced gastric cancer who had failed standard treatment with FGFR1-3 variant, were included in the study by meeting the inclusion criteria after completing the informed consent. Patients will receive pemitinib 13.5 mg once daily (QD) orally on a 2-week dose / 1-week withdrawal regimen. Subjects will continue treatment until disease progression or intolerable toxicity. Clinical tumor imaging evaluation per RECIST v1.1, every 6 weeks (± 7 days) and every 9 weeks (± 7 days) after 48 weeks. Safety assessment was performed using NCI-CTCAE 5.0.

Pemitinib, dose and mode of administration:

Pemitinib will be treated as a 2 week / 1 week withdrawal regimen, 1 dose, 13.5mg, QD, 21 day cycle. Subjects should be on pometitinib at a fixed time per day to avoid inconsistent effects on plasma concentration.

Sample size and statistical methods:

1. In this study, using the 6-month PFS rate as the primary endpoint, Calculted using the confidence interval method of Kapian-Meier estimation, Based on the historical data, The 6-month PFS rate of second-line chemotherapy in subjects with previous first-line treatment was approximately 20% (RAINBOW study, BRIGHTER Study), The 6-month PFS rate in subjects with previous second-line or more treatment was approximately 10% (Attraction-2 study), It is estimated that about 20% of the second-line and above treated subjects will be included in this study, The overall 6-month PFS rate was about 18%, Assuming that the 6-month PFS rate could be improved to 36%, Using the test level as one-sided α =0.1, ß=0.20, After follow-up for at least 6 months, With 80% confidence be observed with a 90% confidence interval lower bound greater than 18%, In total, 23 subjects will need to be enrolled.
2. Statistical analysis method: Continuous variables were described by mean, standard deviation, median, minimum and maximum values, and categorical variables were described by frequency and percentage. The proportion of subjects with the ORR and DCR and their 95% CI were estimated. Median PFS, DOR, and OS were estimated using Kaplan-Meier.

ELIGIBILITY:
Inclusion Criteria:

-

Main selection criteria:

Written informed consent was signed prior to the implementation of any trial-related process;

1. Age: 18 years old;
2. Advanced gastric cancer was confirmed histologically or cytologically;
3. At least one measurable lesion as per version RECIST v1.1;
4. Histology confirmed the presence of the FGFR1-3 variant, including but not limited to amplification, mutation, fusion / rearrangement;
5. Patients who are tested negative for HER 2 by immunohistochemistry (IHC), or by immunohistochemistry (ICH) and in situ hybridization (ISH);
6. Progressive disease after standard treatment;
7. No previous small molecule multitarget inhibitors containing FGFR pathway (including but not limited to allotinib, lemavatinib, sorafenib, apatinib, etc.);
8. The ECOG physical fitness status is 0-1;
9. Expected survival time of> 3 months;

Exclusion Criteria:

- Written informed consent was signed prior to the implementation of any trial-related process;

1. Age: 18 years old;
2. Advanced gastric cancer was confirmed histologically or cytologically;
3. At least one measurable lesion as per version RECIST v1.1;
4. Histology confirmed the presence of the FGFR1-3 variant, including but not limited to amplification, mutation, fusion / rearrangement;
5. Patients who are tested negative for HER 2 by immunohistochemistry (IHC), or by immunohistochemistry (ICH) and in situ hybridization (ISH);
6. Progressive disease after standard treatment;
7. No previous small molecule multitarget inhibitors containing FGFR pathway (including but not limited to allotinib, lemavatinib, sorafenib, apatinib, etc.);
8. The ECOG physical fitness status is 0-1;
9. Expected survival time of> 3 months;
10. For icient organ function for the following laboratory indicators:

    1. In the absence of granulocyte colony-stimulating factor for the last 14 days (ANC)≥1.5x109/L；
    2. In the last 14 days without blood transfusion, platelets 100109/L；
    3. Hemoglobin> 9 g/dL without blood transfusion or erythropoietin in the last 14 days;
    4. Total bilirubin 1.5 upper limit of normal (ULN); or total bilirubin> ULN but direct bilirubin ULN;
    5. Asparpartate aminotransferase (AST), alanine transaminotransferase (ALT) at 2.5 ULN (ALT or AST 5 ULN is allowed in patients with liver metastasis);
    6. Blood creatinine of 1.5 ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) of 50 ml / min;
    7. The coagulation function is good, defined as the international normalized ratio (INR) or prothrombin time (PT) 1.5 times ULN; if the subject is undergoing anticoagulant therapy, as long as the PT is within the proposed range of the anticoagulant
11. For female subjects of childbearing age, a urine or serum pregnancy test within 3 days prior to the first dose of study drug (cycle 1 Day 1, was negative). If the urine pregnancy test results cannot be confirmed as negative, a blood pregnancy test is required. Non-childbearing women were defined as at least 1 year after menopause, or had undergone surgical sterilization or hysterectomy;
12. If there is a risk of conception, all subjects (either male or female) should have an annual failure rate below 1% for the entire treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy drug).

Main exclusion criteria:

1. Other malignant diseases other than digestive tract tumors diagnosed within 5 years before the first dose (excluding radical skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or radical resection);
2. Previous selective FGFR inhibitor therapy;
3. Have received any other study drug or attended an interventional clinical investigator within 28 days prior to the first dose; or had received antitumor treatment (including herbal medicine with anti-tumor indications) within 28 days prior to the initial dose of the study drug;
4. Not yet adequate recovery from toxicity and / or complications due to any intervention (i. e., grade 1 or at baseline, excluding fatigue or alopecia);
5. Known to of symptomatic CNS metastases and / or cancerous meningitis. The previously treated subjects could participate in the trial if stable (no evidence of radiographic progression within at least 4 weeks before the first dose of trial treatment), repeat imaging confirmed no evidence of new brain metastases or enlargement of lesions, and no steroid treatment was required at least 14 days before the first dose. This exception does not include cancerous meningitis, which should be ruled out regardless of its stable clinical status;
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
7. The following laboratory parameters are abnormal:

   1. Serum phosphates> ULN;
   2. Serum calcium exceeds the normal range, or when serum albumin is beyond the normal range, the corrected calcium concentration of serum albumin is beyond the normal range;
   3. Potassium level <lower normal; potassium level can be corrected by supplements at screening.
8. Known history of human immunodeficiency virus (HIV) infection or confirmed positive immune test results;
9. Severe infection with active period or poor clinical control;
10. Thorachydrate, ascites or pericardial effusion with obvious clinical symptoms and requiring drainage;
11. Patients infected with acute or chronic active hepatitis B or hepatitis C, hepatitis B virus (HBV) DNA> 2000 IU / ml or 104Copy / ml; hepatitis C virus (HCV) RNA> 103Copy / ml; hepatitis B surface antigen (HbsAg) was positive with anti-HCV antibody. After the nucleotide antiviral treatment is lower than the above standards, they can be enrolled;
12. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months before the first dose, New York Heart Association grade III / IV congestive heart failure, and uncontrolled cardiac disorders (allowing pacemaker wear or subjects with atrial fibrillation with good heart rate control);
13. With ECG change or medical history considered clinically significant by the investigator; screen QTcF interval> 480 ms, for subjects with indoor block (QRS interval> 120 ms), use JTc interval instead of QTc interval (if JTc is used instead of QTc, JTc must be 340 ms);
14. Uncontrolled hypertension, systolic blood pressure> 160 mmHg or diastolic blood pressure> 100 mmHg after optimal medical treatment, a history of hypertensive crisis or hypertensive encephalopathy;

Main exclusion criteria:

1. Other malignant diseases other than digestive tract tumors diagnosed within 5 years before the first dose (excluding radical skin basal cell carcinoma, skin squamous epithelial carcinoma, and / or radical resection);
2. Previous selective FGFR inhibitor therapy;
3. Have received any other study drug or attended an interventional clinical investigator within 28 days prior to the first dose; or had received antitumor treatment (including herbal medicine with anti-tumor indications) within 28 days prior to the initial dose of the study drug;
4. Not yet adequate recovery from toxicity and / or complications due to any intervention (i. e., grade 1 or at baseline, excluding fatigue or alopecia);
5. Known to of symptomatic CNS metastases and / or cancerous meningitis. The previously treated subjects could participate in the trial if stable (no evidence of radiographic progression within at least 4 weeks before the first dose of trial treatment), repeat imaging confirmed no evidence of new brain metastases or enlargement of lesions, and no steroid treatment was required at least 14 days before the first dose. This exception does not include cancerous meningitis, which should be ruled out regardless of its stable clinical status;
6. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
7. The following laboratory parameters are abnormal:

   1. Serum phosphates> ULN;
   2. Serum calcium exceeds the normal range, or when serum albumin is beyond the normal range, the corrected calcium concentration of serum albumin is beyond the normal range;
   3. Potassium level <lower normal; potassium level can be corrected by supplements at screening.
8. Known history of human immunodeficiency virus (HIV) infection or confirmed positive immune test results;
9. Severe infection with active period or poor clinical control;
10. Thorachydrate, ascites or pericardial effusion with obvious clinical symptoms and requiring drainage;
11. Patients infected with acute or chronic active hepatitis B or hepatitis C, hepatitis B virus (HBV) DNA> 2000 IU / ml or 104Copy / ml; hepatitis C virus (HCV) RNA> 103Copy / ml; hepatitis B surface antigen (HbsAg) was positive with anti-HCV antibody. After the nucleotide antiviral treatment is lower than the above standards, they can be enrolled;
12. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months before the first dose, New York Heart Association grade III / IV congestive heart failure, and uncontrolled cardiac disorders (allowing pacemaker wear or subjects with atrial fibrillation with good heart rate control);
13. With ECG change or medical history considered clinically significant by the investigator; screen QTcF interval> 480 ms, for subjects with indoor block (QRS interval> 120 ms), use JTc interval instead of QTc interval (if JTc is used instead of QTc, JTc must be 340 ms);
14. Uncontrolled hypertension, systolic blood pressure> 160 mmHg or diastolic blood pressure> 100 mmHg after optimal medical treatment, a history of hypertensive crisis or hypertensive encephalopathy;
15. Hepatic encephalopathy, hepatorenal syndrome or Child-Pugh B or more severe cirrhosis.
16. A major surgical procedure (craniotomy, thoracotomy or laparotomy) within 4 weeks prior to the first dose of study treatment or is expected to require major surgery during the study treatment;
17. Complications of toxicity and / or major surgery have not recovered sufficiently before starting treatment;
18. Women in pregnancy or lactating, or subjects expected to be pregnant or born during the study from the screening visit to completion of the safety follow-up visit (male subjects to 90 days after the last dose);
19. Received radiotherapy within 4 weeks before the first dose of the study drug. The subject with radiotherapy-related toxicity must have fully recovered and not require corticosteroid therapy, confirming the exclusion of radiation pneumonia. For palliative radiotherapy for non-CNS disease, a 2-week washout period is allowed;
20. A history of systemic electrolyte metabolic imbalance with calcium and phosphorus metabolism disorders or soft tissue ectopic calcification (except for the calcification of skin, kidney, tendon, or vascular soft tissue without systemic electrolyte metabolic imbalance caused by injury, disease, and advanced age);
21. Clinically significant corneal or retinal disease confirmed by ophthalmic examination;
22. Any potent CYP3A4 inhibitor (see Appendix A) or inducer has been used for 14 days or 5 half-lives (whichever shorter) prior to the first dose of the study drug. Exogenous use of ketoconazole is allowed;
23. Known allergic reactions to peometinib or peometinib study drug excipients;
24. Failure or unwillingness to swallow peimitinib or significant digestive diseases that may interfere with absorption, metabolism or excretion;
25. The subject had a history of vitamin D deficiency and needed an excessive amount of vitamin D supplementation (except for vitamin D dietary supplements);
26. Other acute or chronic illness, mental illness, or abnormal laboratory tests that may increase the risk of study participation or study drug administration or interfere with the interpretation of study results and identify the patient as ineligible for the study in the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 23 (Estimated)
Dates: Start 2023-08-25 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
PFS | 6-month PFS
  to evaluate the efficacy of pemitinib in patients with advanced gastric cancer who have previously failed standard therapy with FGFR1-3 variants

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer center of SunYat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No